CLINICAL TRIAL: NCT02156453
Title: The Evaluation of Short-term Functional Recovery of Total Knee Arthroplasty Patients
Brief Title: Functional Recovery After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 126/2556(EC2)
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Knee Osteoarthritis
Keywords: Functional recovery; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total knee arthroplasty: Patients undergoing uncomplicated total knee replacement
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — All patients will undergo total knee replacement using midvastus approach by single surgeon.

SUMMARY:
Total knee replacement is one of the most successful surgical procedures in Orthopaedics. However, 10-20% of the patients are still dissatisfied with the results of the surgery. In general, the evaluation of postoperative functional outcomes are usually measured by self-report questionnaires, such as the Western Ontario and Mcmaster Universities osteoarthritic Index (WOMAC) and the Short Form-36 health survey (SF-36). Another method to evaluate functional outcome of the patients is to use the performance-based tests such as the two-minute walk test, but there is still little information regarding its use for evaluating functional recovery in patients receiving total knee arthroplasty.

The objectives this study are: 1) to assess the relationship between self-report questionnaires and performance-based tests among patients scheduling for TKA; and 2) to identify clinical variables that are associated with pre- and postoperative functional performance of the patients.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is one of the most prevalent age-related musculoskeletal conditions, resulting in significant impairment in patients' abilities to perform activities and adversely impacting their quality of life. The level of impairment in patients with knee OA can be measured using validated self-report questionnaires, such as the disease-specific Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the generic Medical Outcomes Study Short Form-36 (SF-36). Self-report questionnaires have been recommended by some investigators for their high internal consistency and ease of administration. Another method to evaluate physical function in patients with knee OA is to use performance-based tests. These tests are tools that assess patients' ability to execute a task in a standardized environment, and include the 2-minute walk test (2MWT) and the timed get-up-and-go test (TUG).

Among all the self-reported questionnaires for knee OA, the WOMAC is one of the most commonly used for baseline assessment and for measurement of treatment outcome, and has been validated for patients undergoing total knee arthroplasty (TKA). Although the WOMAC provides information on how individuals perceive their physical function in their own environment, it does not describe their ability to perform a specific task or action. In addition, some investigators showed that scores from self-report questionnaires before and after arthroplasty can overestimate patients' actual functional capacity. For example, Parent et al demonstrated that total knee arthroplasty patients had a dramatic improvement at 2 months as assessed by the WOMAC function subscale, however there were no significant changes when measured with performance-based tests assessing gait speed and stair ascent duration. Therefore, clinicians should be cautious when interpreting findings from studies that provide only self-report questionnaire scores. Given that self-report questionnaires may over-estimate functional status after joint replacement, some authors advocate performance-based tests as measures of outcome, and recommend their use during the preoperative period as baseline measurements followed by subsequent comparison with postoperative measurements.

The objectives of this study are: 1) to assess the relationship between self-reported questionnaires (WOMAC and SF-36) and performance-based tests (2MWT, TUG) among patients scheduling for TKA; and 2) to identify clinical variables that are associated with pre- and post-operative performance of the 2MWT and TUG. Our hypothesis is that correlations between self-report questionnaires and performance-based tests would be low to moderate, and thus these two types of measurements evaluate distinct domains of functional status in patients undergoing TKA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who aged between 40-100 years
* Patients who diagnosed with end-stage osteoarthritis of the knee

Exclusion Criteria:

* Patients who receive total knee replacement on the contralateral side during the past 6 months
* Patients with diseases or conditions that may affect postoperative functional recovery such as severe cardiopulmonary disease
* Unable to participate in postoperative follow-up visits
* Prior surgery on the affected knee, such as high tibial osteotomy
* Patients with complex deformity who require bone grafting or metal augments

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive uncomplicated total knee replacement by a single surgeon
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change of the 2-minute walk test (2MWT) from baseline to at 1 year after surgery | baseline, 6 weeks, 3 months, 6 months and 1 year after surgery

SECONDARY OUTCOMES:
Change of the Timed get-up-and-go test (TUG) from baseline to 1 year after surgery | baseline, 6 weeks, 3 months, 6 months and 1 year after surgery
Change of the pain scores on the Visual Analog Scale from baseline to 1 year after surgery | baseline, 6 weeks, 3 months, 6 months and 1 year after surgery
Change of the functional scores on the WOMAC index (Thai version) from baseline to 1 year after surgery | baseline, 3 months, 6 months and 1 year after surgery
Change of the physical function domain of the SF-36 Health Survey from baseline to 1 year after surgery | baseline, 3 months, 6 months and 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aasis Unnanuntana, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand